CLINICAL TRIAL: NCT02886130
Title: Effects of Alpha-glycerylphosphorylcholine on Physical and Cognitive Performances in Varsity Volleyball Players
Brief Title: Alpha-GPC and Physical and Cognitive Performances in Volleyball Players.
Acronym: VolleyAGPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Raynald Bergeron, Associate professor, Université de Montréal
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Montreal
Record Dates: First submitted 2016-08-24; First posted 2016-09-01 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Athletic Performance
Keywords: Alpha-GPC; Volleyball; Athletes; Executive functions; Vertical jump; Peak power
MeSH Terms: interventions — maltodextrin; Glycerylphosphorylcholine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Maltodextrin tablets (4x per day) 2 x 250 mg in the morning, 2 x 250 mg 60 min before workout, 4 weeks duration
  Interventions: Dietary Supplement: Placebo
- Alpha-GPC (Experimental): Alpha-GPC tablets (4x per day) 2 x 250 mg in the morning, 2 x 250 mg 60 min before workout, 4 weeks duration
  Interventions: Dietary Supplement: Experimental

INTERVENTIONS:
Dietary Supplement: Placebo — Monitoring of supplementation (e.g., compliance, subject blindness), diet (to control dietary choline ingestion), training volume and adverse effects will be performed on a weekly basis to ensure maximal control of confounding factors as well as the safety of volunteers during the study.
  Other Names: Maltodextrin; Control
  Arms: Placebo
Dietary Supplement: Experimental — Monitoring of supplementation (e.g., compliance, subject blindness), diet (to control dietary choline ingestion), training volume and adverse effects will be performed on a weekly basis to ensure maximal control of confounding factors as well as the safety of volunteers during the study.
  Other Names: Alpha-gpc; Alpha-glycerylphosphorylcholine; Alpha-gpc supplementation; A-GPC
  Arms: Alpha-GPC

SUMMARY:
In order to attain the elite level on the national scene, volleyball players need several attributes. In addition to mastering technical and tactical skills, great jumping ability is another important asset. Maximal power output needed to achieve height during a jump necessitates coordinated neuromuscular recruitment and muscle mass among others. Interestingly, there are claims that alpha-glycerylphosphorylcholine (A-GPC) increases acetylcholine synthesis and enhances exercise-induced increases in plasma growth hormone concentrations, two factors that could theoretically be associated neuromuscular transmission and muscle mass.

However, until now only a few studies have investigated the role of A-GPC in human exercise performance. Published results were mixed. One recent study showed that isometric peak force was slightly but significantly increased when subjects had ingested a daily dose of 600 mg of A-GPC over a period of 6 days (Bellar et al., JISSN, 2015).

The objective of our study is to evaluate the longer-term effects (4 weeks) using a higher dose (1000 mg/day) of A-GPC on jumping capabilities in elite male and female volleyball players.

DETAILED DESCRIPTION:
Our study design will be a placebo controlled, randomized, double-blind, crossover study. Varsity male and female volleyball players (n=28) will each be asked to participate in both arms of the study, i.e. placebo and A-GPC (1000 mg/kg/day). The duration of each arm of the study will be 4 weeks separated by a 7-day washout period. The order of treatment (placebo or A-GPC) will be determined randomly. Athletes will be asked to maintain their training load during the duration of the experiment.

ELIGIBILITY:
Inclusion Criteria:

* Be a competitive varsity volleyball player

Exclusion Criteria:

* Regular consumption of alpha-GPC within the last 4 months
* Receiving drug treatment except 1) contraception (pill), and 2) treatment against asthma

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2016-12-20 (Actual); Study Completion 2016-12-20 (Actual)

PRIMARY OUTCOMES:
Change in countermovement jump performance at 4 weeks | Assessments at week 0 and at week 4 of supplementation or placebo
  Jump height is calculated using two forces plates which measures the time the feet are off the platform. The athlete stands upright with weight evenly distributed over both feet. Hands are placed on the hips, and stay there throughout the test. When all is ready, the athlete squats down until the knees are bent at 90 degrees, then immediately jumps vertically as high as possible, landing back on the platform on both feet at the same time. Allow a good rest between trials. The take-off must be from both feet, with no initial steps or shuffling. They must also not pause at the base of the squat.

SECONDARY OUTCOMES:
Change in vertical jump - run up at 4 weeks | Assessments at week 0 and at week 4 of supplementation or placebo
  Record the standing height of the subject by getting then to stand directly below the apparatus with both feet on tip-toes, and then stretch up one arm and reach as high as possible. The subject then stands the appropriate distance from the base of the apparatus (about 15 feet), and when ready take 3 or so steps before leaping off up off both legs as high as possible, using the arms to assist in projecting the body upwards. The subject should aim to take off just short of the apparatus, so that at the peak of the jump they are directly under it.
Executive function | After 4 weeks of supplementation or placebo
  "Task switching" is a useful tool to investigate executive functions in humans. This task allows investigation of the ability to maintain, select and switch among task sets.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel St-Arnaud, B.Sc, Principal Investigator — Université de Montréal; Raynald Bergeron, Ph.D, Study Director — Université de Montréal; Jonathan Tremblay, Ph.D, Study Director — Université de Montréal
Locations (1):
- CEPSUM (Centre d'éducation physique et des sports de l'université de Montréal), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual data obtained from vertical jump assessments and during the cognitive switch task will be communicated to each athlete.

REFERENCES:
- [Background] Bellar D, LeBlanc NR, Campbell B. The effect of 6 days of alpha glycerylphosphorylcholine on isometric strength. J Int Soc Sports Nutr. 2015 Nov 17;12:42. doi: 10.1186/s12970-015-0103-x. eCollection 2015. PMID 26582972
- [Background] Barbagallo Sangiorgi G, Barbagallo M, Giordano M, Meli M, Panzarasa R. alpha-Glycerophosphocholine in the mental recovery of cerebral ischemic attacks. An Italian multicenter clinical trial. Ann N Y Acad Sci. 1994 Jun 30;717:253-69. doi: 10.1111/j.1749-6632.1994.tb12095.x. PMID 8030842
- [Background] Hoffman JR, Ratamess NA, Gonzalez A, Beller NA, Hoffman MW, Olson M, Purpura M, Jager R. The effects of acute and prolonged CRAM supplementation on reaction time and subjective measures of focus and alertness in healthy college students. J Int Soc Sports Nutr. 2010 Dec 15;7:39. doi: 10.1186/1550-2783-7-39. PMID 21156078
- [Background] Kidd PM. Integrated brain restoration after ischemic stroke--medical management, risk factors, nutrients, and other interventions for managing inflammation and enhancing brain plasticity. Altern Med Rev. 2009 Mar;14(1):14-35. PMID 19364191
- [Background] Parnetti L, Amenta F, Gallai V. Choline alphoscerate in cognitive decline and in acute cerebrovascular disease: an analysis of published clinical data. Mech Ageing Dev. 2001 Nov;122(16):2041-55. doi: 10.1016/s0047-6374(01)00312-8. PMID 11589921
- [Background] Traini E, Bramanti V, Amenta F. Choline alphoscerate (alpha-glyceryl-phosphoryl-choline) an old choline- containing phospholipid with a still interesting profile as cognition enhancing agent. Curr Alzheimer Res. 2013 Dec;10(10):1070-9. doi: 10.2174/15672050113106660173. PMID 24156263
- [Background] Zeisel SH. A brief history of choline. Ann Nutr Metab. 2012;61(3):254-8. doi: 10.1159/000343120. Epub 2012 Nov 26. PMID 23183298
- [Background] Gajewski PD, Wild-Wall N, Schapkin SA, Erdmann U, Freude G, Falkenstein M. Effects of aging and job demands on cognitive flexibility assessed by task switching. Biol Psychol. 2010 Oct;85(2):187-99. doi: 10.1016/j.biopsycho.2010.06.009. Epub 2010 Jul 3. PMID 20599468
- See also: The effects of alpha-glycerylphosphorylcholine, caffeine or placebo on markers of mood, cognitive function, power, speed, and agility — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4595381/